CLINICAL TRIAL: NCT03086538
Title: Pemetrexed Plus Tarceva as Salvage Treatment in EGFR Overexpressed Metastatic Colorectal Cancer Patients Who Were Failed After Standard Chemotherapy: A Phase II Single Arm Prospective Study
Brief Title: Pemetrexed Plus Tarceva as Salvage Treatment in EGFR Overexpressed Metastatic Colorectal Cancer Patients Who Were Failed After Standard Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-046
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Pemetrexed; Erlotinib Hydrochloride; Tablets

STUDY DESIGN:
Intervention Model Description: Pemetrexed 500 mg/m2 IV Q 3 weeks Tarceva 100mg once daily, continous
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pemetrexed+Tarceva (Experimental): Pemetrexed 500 mg/m2 IV Q 3 weeks Tarceva 100mg once daily, continous
  Interventions: Drug: Pemetrexed; Drug: Tarceva 100Mg Tablet

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed is a multitarget antifolate (MTA) whose mechanism of action relies mainly on the inhibition of TS, with weaker secondary effects on glycinamide ribonucleotide formyltransferase (GARFT) and dihydrofolate reductase (DHFR), leading to impairment of DNA synthesis and repair.
Drug: Tarceva 100Mg Tablet — Erlotinib (tarceva) is oral epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI).

SUMMARY:
This study is single center single arm prospective phase II study. In this study, efficacy and side effects of pemetrexed as salvage regimen on patients who failed all standard chemotherapy and total of 29 patients will be enrolled. Pemetrexed will be continued until disease progression is happened.

DETAILED DESCRIPTION:
Antitumor effect of pemetrexed is already proven lung cancer, pleural mesothelioma, peritoneal mesothelioma and has been used as a standard therapeutic agent. In addition, this drug does not have severe side effects, pemetrexed is thought to be an important option for patients with poor performance status or elderly patients. Pemetrexed has been studied in colorectal cancer, Zhang et al have demonstrated that pemetrexed combined with gefitinib has a significantly synergistic effect on colorectal cancer cells (17). In two phase II studies in which patients received pemetrexed as first-line treatment for metastatic disease, objective response rates were 15 - 17 %. These trials were conducted prior to supplementation with folic acid and vitamin B12, which markedly decreased the frequency of hematologic toxicities of pemetrexed; routine supplementation is now included in all clinical trials of the agent (18).

Erlotinib (tarceva) is oral epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI). Erlotinib showed the effect in the maintanence therapy (combined with bevacizumab) in colorector cancer. Also, erolitinib had the effect in biliary tract cancer and pancreatic cancer. Our previous phase III trial for tarceva puls GEMOX (gemcitabine plus oxaliplatin) reported that adding to tarceva to GEMOX had more useful in the specific subgroup with EFGR overexpressed patients.

The aim of present study is to assess treatment efficacy and side effects of pemetrexed plus tarceva on EGFR overexpressed patients with refractory colorectal cancer and no treatment option whose performance status is relatively preserved.

<Pre-medication for Alimta> D-7 ~ Folic acid 1mg QD PO D-7 ~ Vitamin B12 1mg/9weeks IM D-1, D1, D2 Dexamethasone 4mg BID PO

<Treatment> D1 Alimta 500mg/m2 + NS 100ml IV infusion for 10mins Every 3weeks

ELIGIBILITY:
Inclusion Criteria:

* Advanced colorectal cancer failed from all standard chemotherapy

  * History of refractoriness from chemotherapy including 5-FU, Oxaliplatin, Irinotecan
  * Oral 5-FU agents are included standard chemotherapy
  * Targeted agents such as cetuximab or bevacizumab are not included in inclusion criteria
* Patient must have willingness and ability to comply with the study protocol including visiting hospital for test and treatment during trial
* ECOG performance status 0~2
* Measurable lesion (RECIST 1.1) must exist
* Expected survival should be more than 3 months from first dose of pemetrexed
* Adequate organ function as defined as below estimated 28 days before first doe of pemetrexed:

Exclusion Criteria:

* Poor performance status (ECOG PS ≥ 3)
* Patient can not take folic acid or Vitamin B12.
* History of previous treatment with pemetrexed
* History of malignant disease, except: non-melanoma skin cancer that properly treated, cured uterine cervical cancer or other solid tumor without evidence of recurrence within 5 years
* Patient can not swallow oral pills.
* Treatment with medication of clinical trial within 14 days (or longer duration according to specific agents)
* Systemic chemotherapy or radiation (except palliative purpose) within 3 weeks (or longer duration according to specific agents)
* Toxicity from previous treatment as CTCAE grade > 1, except alopecia
* bowel obstruction or CTCAE grade 3/4 upper GI bleeding before 4 weeks
* QTc prolongation (QTc > 480msec) at resting is documented more than twice within 24 hours or family history of QT prolongation syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Hong JY, Lee J, Park JO, Lim HY, Kang WK, Park YS. Pemetrexed/Erlotinib as a Salvage Treatment in Patients with High EGFR-Expressing Metastatic Colorectal Cancer Following Failure of Standard Chemotherapy: A Phase II Single-Arm Prospective Study. Target Oncol. 2020 Feb;15(1):67-73. doi: 10.1007/s11523-019-00691-z. PMID 31820199